CLINICAL TRIAL: NCT02214862
Title: Pilot, Exploratory Study With [F18]-FDDNP-PET for in Vivo Diagnose of Tauopathy in Unclassified Parkinsonism
Brief Title: 2-(1-{6-[(2-[F-18]Fluoroethyl) (Methyl)Amino]-2-naphthyl} Ethylidene) Malononitrile-PET for in Vivo Diagnose of Tauopathy in Unclassified Parkinsonism
Acronym: [F18]-FDDNP
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Fundacion Clinic per a la Recerca Biomédica (Other)
Responsible Party: Principal Investigator, Maria Jose Martí, MD, PhD, Fundacion Clinic per a la Recerca Biomédica
Allocation: Not Applicable | Model: Single Group | Masking: None
Other Study IDs: PI11/02031
Record Dates: First submitted 2014-08-11; First posted 2014-08-12 (Estimated); Last update posted 2016-02-04 (Estimated); Status verified 2016-02

CONDITIONS: Progressive Supranuclear Palsy; Multi-System Atrophy; Parkinsonism
Keywords: Unclassifiable Parkinsonism, [F18]-FDDNP-PET, Tauopathy, PSP,MSA
MeSH Terms: conditions — Supranuclear Palsy, Progressive; Parkinsonian Disorders; Tauopathies | interventions — dicyanmethane

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- [F18]-FDDNP (Experimental): 2-(1-{6-[(2-[F-18]fluoroethyl) (methyl)amino]-2-naphthyl} ethylidene) malononitrile Radiopharmaceutical tracer, intravenous, single dose of 360+/-20 megabecquerel
  Interventions: Drug: [F18]-FDDNP

INTERVENTIONS:
Drug: [F18]-FDDNP — radiopharmaceutical tracer
  Other Names: 22-(1-{6-[(2-[F-18]fluoroethyl) (methyl)amino]-2-naphthyl} ethylidene) malononitrile

SUMMARY:
The PET tracer [F18]-FDDNP has a specific affinity for lesions containing tau protein.

The study consists of two phases:

* In the first (cross-sectional) phase it will be assessed the uptake of [18F]-FDDNP in 10 cases with progressive supranuclear palsy (PSP, a tauopathy) en 10 with multi-system atrophy (MSA, a non-tauopathy), along with 20 individuals with Unclassifiable Parkinsonism, as previously defined in a European cohort study.
* In the second (longitudinal) phase it will be prospectively followed the 20 unclassifiable patients (at 6, 12 and 18 months) by means of validated scales and accepted diagnostic criteria in order to try to correlate their eventual clinical diagnosis with baseline PET findings. On this basis, we endeavour to estimate the ability of this technique to detect in vivo underlying tau pathology in subjects initially unclassifiable on clinical grounds.

We hypothesized that:

1. Patients with clinically definite PSP will present an increased uptake in basal ganglia, brainstem and cerebellum.
2. Patients with clinically defined MSA will not present specific uptake.
3. Part of unclassifiable patients with parkinsonism will present a pattern of uptake similar to patients with clinically defined PSP and this part along the clinical follow-up will be meet clinical criteria for diagnose of PSP

ELIGIBILITY:
Inclusion Criteria:

* The subject is male or female ≥ 40 years old;
* The individual has one of these three conditions:
* probable PSP according to criteria of the National Institute of Neurological Disorders and Stroke (NINDS)
* probable MSA according to criteria of the Second consensus statement on the diagnosis of multiple system atrophy
* unclassifiable parkinsonism according to criteria defined by Katzenschlager et al, 2003:
* Patients with atypical parkinsonism without response to treatment with levodopa and does not meet any of the diagnostic criteria for other known atypical parkinsonism
* Patient given written consent

Exclusion Criteria:

* The subject is diagnosed with Parkinson's Disease and meets the diagnostic criteria United Kingdom Parkinson's Disease Society Brain Bank -The subject is pregnant or breastfeeding;
* The subject has a history of drug abuse or alcohol;
* The subject has a moderate or severe renal function impairment (creatinine serum> 1.5 mg / dL);
* The subject has a moderate or severe hepatic impairment (bilirubin> 2 times the upper limit of normal, transaminases> 3 times the limit top of normal);
* The subject presents structural abnormalities in the basal ganglia or cortical level on MRI or CT;
* The subject has participated in a clinical study with a pharmaceutical product investigation within 30 days prior to screening and / or a radiopharmaceutical minimum period of 5 radioactive half-lives prior to screening;
* Occupational exposure to radiation> 15 milliSievert (mSv) / year
* Use of nonsteroidal antiinflammatory drug (NSAIDs), for some reason, can not be replaced by any other drug 4 weeks before the PET scan;
* The subject has allergy investigational product or any of its components;
* The subject has a clinically severe active disease, with a hope reduced life;
* The subject is claustrophobic / a.

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2013-03; Primary Completion 2015-12 (Actual); Study Completion 2016-02 (Actual)

PRIMARY OUTCOMES:
To assess the Relative Volume of Distribution of [18F]-FDDNP in individuals with unclassifiable parkinsonism, and to try to correlate their eventual clinical diagnosis with baseline PET findings. | 18 months

SECONDARY OUTCOMES:
to assess the uptake of [18F]-FDDNP in cases clinically defined of progressive supranuclear palsy and multi-system atrophy | Baseline assessment
To assess the ability to detect in vivo underlying tau pathology in unclassifiable parkinsonism by means of PET -[18F]-FDDNP. | 18 months

CONTACTS AND LOCATIONS:
Overall Officials: Maria Jose Martí, Md, PhD, Principal Investigator — Fundació per a la Recerca Biomedica
Locations (1):
- Hospital Clinic, Barcelona, Spain, Spain

REFERENCES:
- [Background] Katzenschlager R, Cardozo A, Avila Cobo MR, Tolosa E, Lees AJ. Unclassifiable parkinsonism in two European tertiary referral centres for movement disorders. Mov Disord. 2003 Oct;18(10):1123-31. doi: 10.1002/mds.10523. PMID 14534915
- [Background] Litvan I, Bhatia KP, Burn DJ, Goetz CG, Lang AE, McKeith I, Quinn N, Sethi KD, Shults C, Wenning GK; Movement Disorders Society Scientific Issues Committee. Movement Disorders Society Scientific Issues Committee report: SIC Task Force appraisal of clinical diagnostic criteria for Parkinsonian disorders. Mov Disord. 2003 May;18(5):467-86. doi: 10.1002/mds.10459. PMID 12722160
- [Background] Gilman S, Wenning GK, Low PA, Brooks DJ, Mathias CJ, Trojanowski JQ, Wood NW, Colosimo C, Durr A, Fowler CJ, Kaufmann H, Klockgether T, Lees A, Poewe W, Quinn N, Revesz T, Robertson D, Sandroni P, Seppi K, Vidailhet M. Second consensus statement on the diagnosis of multiple system atrophy. Neurology. 2008 Aug 26;71(9):670-6. doi: 10.1212/01.wnl.0000324625.00404.15. PMID 18725592
- [Background] Golbe LI, Ohman-Strickland PA. A clinical rating scale for progressive supranuclear palsy. Brain. 2007 Jun;130(Pt 6):1552-65. doi: 10.1093/brain/awm032. Epub 2007 Apr 2. PMID 17405767
- [Background] Wenning GK, Tison F, Seppi K, Sampaio C, Diem A, Yekhlef F, Ghorayeb I, Ory F, Galitzky M, Scaravilli T, Bozi M, Colosimo C, Gilman S, Shults CW, Quinn NP, Rascol O, Poewe W; Multiple System Atrophy Study Group. Development and validation of the Unified Multiple System Atrophy Rating Scale (UMSARS). Mov Disord. 2004 Dec;19(12):1391-402. doi: 10.1002/mds.20255. PMID 15452868
- [Background] Wong KP, Wardak M, Shao W, Dahlbom M, Kepe V, Liu J, Satyamurthy N, Small GW, Barrio JR, Huang SC. Quantitative analysis of [18F]FDDNP PET using subcortical white matter as reference region. Eur J Nucl Med Mol Imaging. 2010 Mar;37(3):575-88. doi: 10.1007/s00259-009-1293-8. Epub 2009 Oct 31. PMID 19882153
- [Background] Buongiorno M, Compta Y, Marti MJ. Amyloid-beta and tau biomarkers in Parkinson's disease-dementia. J Neurol Sci. 2011 Nov 15;310(1-2):25-30. doi: 10.1016/j.jns.2011.06.046. Epub 2011 Jul 20. PMID 21764078
- [Background] Smid LM, Vovko TD, Popovic M, Petric A, Kepe V, Barrio JR, Vidmar G, Bresjanac M. The 2,6-disubstituted naphthalene derivative FDDNP labeling reliably predicts Congo red birefringence of protein deposits in brain sections of selected human neurodegenerative diseases. Brain Pathol. 2006 Apr;16(2):124-30. doi: 10.1111/j.1750-3639.2006.00006.x. PMID 16768752